CLINICAL TRIAL: NCT06361979
Title: A Single-arm, Exploratory Clinical Study of SHR-A1811 Combined With Bevacizumab in the Treatment of HER2-positive Breast Cancer With Brain Metastases
Brief Title: SHR-A1811 Combined With Bevacizumab in HER2-positive Breast Cancer With Brain Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Huihua Xiong (Other)
Responsible Party: Sponsor-Investigator, Huihua Xiong, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1811
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Breasr Cancer
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARM1 (Experimental)
  Interventions: Drug: SHR-A1811; Drug: Bevacizumab

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811: intravenous
Drug: Bevacizumab — Bevacizumab:intravenous

SUMMARY:
This study aimed to evaluate the use of SHR-A1811 and bevacizumab in HER2-positive Breast Cancer with brain metastases

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. Pathologically confirmed HER2-positive breast cancer;
3. At least one measurable intracranial lesion according to RANO-BM criteria, which had not received local treatment;
4. More than 2 weeks from last systemic treatment; patients with new brain lesions after craniocerebral surgery were admitted if no radiotherapy was performed.
5. Prior HER2-target treatment, endocrine therapy and chemotherapy was allowed;
6. Adequate function of major organs-

Exclusion Criteria:

1. Previous treatment with trastuzumab deruxtecan (DS-8201a) or any other antibody drug conjugate (ADC) which consists of an exatecan derivative that is a topoisomerase 1 inhibitor;
2. Previous treatment with bevacizumab;
3. Participated in other drug clinical trials within 4 weeks before admission;
4. History of clinically significant lung disease；
5. Other malignant tumors, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma, have been diagnosed in the past five years.
6. According to the judgement of the researchers, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of research (including, but not limited to, severe hypertension, severe diabetes, active infections, etc.).
7. Any other conditions that researchers believe that patients are unsuitable for this study.

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
CNS-ORR | Up to 2 years
  CNS-ORR was defined as percentage of participants with CNS response assessed by the investigator according to RANO-BM criteria

SECONDARY OUTCOMES:
PFS | up to 2 years
  PFS was defined as the time from first dose to first documented disease progression (PD) or death from any cause, whichever occurred first
ORR | Up to 2 years
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR assessed by the investigator according to RECIST version 1.1
AE | Up to 2 years
  Proportion of participants experienced adverse events during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Xiong huihua, Principal Investigator — Tongji Hospital Affiliated of Tongji Medical College Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: Undecided